CLINICAL TRIAL: NCT01066351
Title: Efficacy of Erythropoietin to Prevent Acute Kidney Injury in Chronic Kidney Disease Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Thammasat University (Other)
Responsible Party: Adis Tasanarong, Faculty of Medicine, Thammasat University (Rangsit Campus)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MTU-E-1-57/52
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-01

CONDITIONS: Acute Renal Failure
Keywords: acute kidney injury; erythropoietin; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — epoetin beta; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Experimental): The patients were assigned to receive beta erythropoietin (Recormon) dose 200 unit/kg at 3 day before cardiac surgery and 100 unit/kg in the morning before cardiac surgery.
  Interventions: Drug: beta erythropoietin
- placebo (Placebo Comparator): The patients were assigned to receive normal saline same volume at 3 day before cardiac surgery and in the morning before cardiac surgery.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: beta erythropoietin — The patients were assigned to receive beta erythropoietin (Recormon) dose 200 unit/kg at 3 day before cardiac surgery and 100 unit/kg in the morning before cardiac surgery.
  Other Names: Recormon
  Arms: Erythropoietin
Drug: placebo — The patients were assigned to receive normal saline same volume at 3 day before cardiac surgery and in the morning before cardiac surgery.
  Other Names: normal saline
  Arms: placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of erythropoietin for prevention acute kidney injury in CKD patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI)occur 7.7-42% after cardiac surgery. The incidence of AKI requiring renal replacement therapy following coronary artery bypass grafting (CABG) surgery was 0.7-3.5% and increase mortality rate. Erythropoietin (EPO) is now considered a novel anti-apoptotic and anti-inflammatory action. The present study was designed to evaluate the administration of EPO as a means of preventing AKI in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years.
* serum creatinine levels > 1.2 mg/dL and baseline creatinine clearance levels < 60 mL/min (as measured in their most recent sample,drawn within 2 months prior to the beginning of the study)
* patients who need cardiac surgery

Exclusion Criteria:

* patients with acute kidney injury
* end stage renal disease (requiring dialysis)
* unstable renal function (as evidenced by a change in serum creatinine of > 0.5 mg/dL, or > 25%, within 14 days prior to the study)
* allergy to any of erythropoietin
* suffered from congestive heart failure, cardiogenic shock or emergent cardiac surgery.
* receiving erythropoietin within 14 days before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-03 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The primary end-point of this study is the development of AKI in placebo group compared with EPO group. | 1.5 year

SECONDARY OUTCOMES:
The secondary end-point of this study is compare urine NGAL level in AKI patients between both groups | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Adis Tasanarong, MD, Principal Investigator — Thammasat Universuty
Locations (1):
- Adis Tasanarong, Khlong Luang, Pathumtani, Thailand

REFERENCES:
- [Background] Song YR, Lee T, You SJ, Chin HJ, Chae DW, Lim C, Park KH, Han S, Kim JH, Na KY. Prevention of acute kidney injury by erythropoietin in patients undergoing coronary artery bypass grafting: a pilot study. Am J Nephrol. 2009;30(3):253-60. doi: 10.1159/000223229. Epub 2009 Jun 2. PMID 19494484
- [Background] Bahlmann FH, Fliser D. Erythropoietin and renoprotection. Curr Opin Nephrol Hypertens. 2009 Jan;18(1):15-20. doi: 10.1097/MNH.0b013e32831a9dde. PMID 19077684
- [Background] Bernhardt WM, Eckardt KU. Physiological basis for the use of erythropoietin in critically ill patients at risk for acute kidney injury. Curr Opin Crit Care. 2008 Dec;14(6):621-6. doi: 10.1097/MCC.0b013e328317ee82. PMID 19005302
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879
- [Derived] Tasanarong A, Duangchana S, Sumransurp S, Homvises B, Satdhabudha O. Prophylaxis with erythropoietin versus placebo reduces acute kidney injury and neutrophil gelatinase-associated lipocalin in patients undergoing cardiac surgery: a randomized, double-blind controlled trial. BMC Nephrol. 2013 Jul 5;14:136. doi: 10.1186/1471-2369-14-136. PMID 23829828
- See also: The Nephrology Society of Thailand — http://www.nephrothai.org/